CLINICAL TRIAL: NCT05858060
Title: Practice of Osmotherapy in Severe SubArachnoid Hemorrhage Patients: Multicenter Observational Study (OSMO-SAH Study)
Brief Title: Osmotic Therapy for Patients With Severe Subarachnoid Hemorrhage
Acronym: OSMO-SAH
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Lidan Jiang, Principal Investigator, Xuanwu Hospital, Beijing
Other Study IDs: XWNeurosurgicalICU
Record Dates: First submitted 2023-05-04; First posted 2023-05-15 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-01

CONDITIONS: Subarachnoid Hemorrhage, Traumatic
Keywords: Subarachnoid Hemorrhage, mannitol, hypertonic saline, outcome
MeSH Terms: conditions — Subarachnoid Hemorrhage, Traumatic; Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — regular blood sample for examination of regular blood chemicals
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this prospective multi-center observational study is to learn about the osmotic therapy in severe subarachnoid hemorrhage (SAH). The main question[s] it aims to answer are:

• whether the two osmotic therapy, 20% mannitol and 10% hypertonic saline(HTS), under the same osmotic equivalent, has similar influence on the outcome of SAH patients?

Participants will be given proper treatment according to local expert consensus, including the choice of osmotic medicine. Investigators just record and analyse the data, compare mannitol group and HTS group to see if the outcome of latter is not worse than the former.

ELIGIBILITY:
Inclusion Criteria:

* ①age ≥18； ②aneurysmal subarachnoid hemorrhage; ③Hunt-Hess 3-5级

Exclusion Criteria:

* previous cranial decompression surgery, cerebrospinal fluid leakage or drainage,

  * bilateral pupils fixed or dilated,

    * hemodynamic instability,

      * hemoglobin < 8g / L,

        * serum osmolality > 320 mOsm / L,

          ⑥ combined with severe organ dysfunction (cardiac, pulmonary, hepatic, renal and so on);

          ⑦ serious electrolyte disorders (serum sodium concentration <125 mmol / L or >170 mmol / L), and difficult to correct within limited time;

          ⑧ serious acid-base balance disorders, and difficult to correct within limited time;

          ⑨ use of mannitol or HSS within previous six hours;

          ⑩ being pregnant.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet inclusion and exclusion criterias will be consecutively included. Treatment will be given according to expert consensus of local center, including neurosurgical and intensive management.
Sampling Method: Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
modified Rankin score | 1 month after ictus
  The Modified Rankin Score (mRS) is the most widely used outcome measure for brain injured patients, which ranges from 0-6. Score of 6 means that patient is dead.
modified Rankin score | 6 months
  The Modified Rankin Score (mRS) is the most widely used outcome measure for brain injured patients, which ranges from 0-6. Score of 6 means that patient is dead.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Jiang L, Qi M, Xu Y, Qu X, Chen W, Cheng W, Zhao H, Shang F, Fu X, Wang C, Jiang R, Wang N. Hyperosmolar therapy for severe subarachnoid haemorrhage: a protocol for a multicentre prospective observational study (OSMO-SAH study). BMJ Open. 2025 Jul 25;15(7):e099008. doi: 10.1136/bmjopen-2025-099008. PMID 40713038